CLINICAL TRIAL: NCT06589986
Title: A Phase III, Multicenter, Double-Blind, Placebo-Controlled, Treat-Through Study to Assess the Efficacy and Safety of Induction and Maintenance Therapy With RO7790121 in Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Assess the Efficacy and Safety of Afimkibart (Also Known as RO7790121) for Induction and Maintenance Therapy in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: Ametrine-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA45329; 2024-513014-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Moderately to Severely Active Ulcerative Colitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Afimkibart (Experimental): Participants will receive afimkibart intravenously (IV) followed by afimkibart subcutaneous (SC) injection.
  Interventions: Drug: Afimkibart
- Placebo (Placebo Comparator): Participants will receive placebo IV followed by placebo SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afimkibart — Afimkibart will be administered as IV infusion. Afimkibart will be administered as SC injection.
  Other Names: PF-06480605; RVT-3101; RG6631; RO7790121
  Arms: Afimkibart
Drug: Placebo — Placebo matching IV afimkibart. Placebo matching SC afimkibart.
  Arms: Placebo

SUMMARY:
This Phase III, multicenter, double-blind, placebo-controlled, treat-through study will evaluate the efficacy and safety of Afimkibart (RO7790121) compared with placebo in participants with moderately to severely active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of UC
* Moderately to severely active UC assessed by mMS
* Bodyweight >= 40 kilogram (kg)
* Up to date with colorectal cancer (CRC) screening performed according to local standards
* Demonstrated inadequate response, loss of response and/or intolerance to at least one protocol-specified conventional or advanced UC therapy
* Males and females of childbearing potential must meet protocol criteria for contraception requirements

Exclusion Criteria:

* Currently known complications of UC (e.g. fulminant colitis, toxic megacolon)
* Current diagnosis of Crohn's disease (CD) or indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis
* Presence of an ostomy or ileoanal pouch
* Current diagnosis or suspicion of primary sclerosing cholangitis
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* Past or current evidence of definite low-grade or high-grade colonic dysplasia or adenomas or neoplasia not completely removed
* History of malignancy within 5 years, with the exception of malignancies adequately treated with resection for non-metastatic basal cell or squamous cell cancer or in situ cervical cancer
* Evidence of infection with Clostridioides difficile (C. difficile; formerly known as Clostridium difficile), cytomegalovirus (CMV), human immunodeficiency virus (HIV), Hepatitis B (HBV), Hepatitis C (HCV)
* Has evidence of active tuberculosis (TB), latent TB not successfully treated (per local guidance) or inadequately treated TB
* Has received protocol-specified prohibited medicines, including known exposure to any type of anti-TL1A therapy

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 12 | At Week 12
  Percentage of participants achieving Modified Mayo Score (mMS) <=2 with stool frequency subscore (SFS) = 0 or 1 (up to 1-2 stools more than normal), rectal bleeding subscore (RBS) = 0 (no blood seen) and endoscopic subscore (ES) = 0 or 1 (normal appearance of mucosa or mild disease) at Week 12. mMS is a composite score of ulcerative colitis disease activity, given by the sum of three subscores: SFS, RBS and ES. Each subscore is measured on a scale from 0 to 3, with higher values associated with greater severity.
Percentage of Participants with Clinical Remission at Week 52 | At Week 52
  Percentage of participants achieving mMS <= 2 with SFS = 0 or 1 (up to 1-2 stools more than normal), RBS = 0 (no blood seen) and ES = 0 or 1 (normal appearance of mucosa or mild disease) at Week 52. mMS is a composite score of ulcerative colitis disease activity, given by the sum of three subscores: SFS, RBS and ES. Each subscore is measured on a scale from 0 to 3, with higher values associated with greater severity.

SECONDARY OUTCOMES:
Change in Partial Modified Mayo Score (pmMS) | Baseline to Week 2
  Change in pmMS from baseline to Week 2. pmMS is a composite score of ulcerative colitis signs and symptoms activity given by the sum of the SFS and RBS. SFS is measured on a scale from 0 (normal number of stools) to 3 (5 or more stools than normal). RBS is measured on a scale from 0 (no blood seen) to 3 (blood alone passed).
Percentage of Participants with Endoscopic Improvement | At Week 12
  Percentage of participants achieving endoscopic subscore of 0 or 1 (normal appearance of mucosa or mild disease) at Week 12.
Percentage of Participants with Endoscopic Remission | At Week 12
  Percentage of participants achieving endoscopic subscore of 0 (normal appearance of mucosa) at Week 12.
Percentage of Participants with Clinical Response | At Week 12
  Percentage of participants achieving a decrease in mMS of at least 2 points and 30% from baseline and either a decrease in RBS >= 1 or RBS = 0 or 1 (no blood seen or stool with streaks of blood) at Week 12. mMS is a composite score of ulcerative colitis disease activity, given by the sum of three subscores: SFS, RBS and ES. SFS is measured on a scale from 0 (normal number of stools) to 3 (5 or more stools than normal). RBS is measured on a scale from 0 (no blood seen) to 3 (blood alone passed). ES is measured on a scale from 0 (normal appearance of mucosa) to 3 (severe disease).
Percentage of Participants with Histologic Improvement | At Week 12
  Percentage of participants achieving a histologic improvement, defined as Geboes <=3.1 at Week 12. Geboes is a grading system for histologic ulcerative colitis disease activity with scores ranging from 0 (no activity) to 5.4 (ulcer or granulation tissue).
Percentage of Participants with Histologic Remission | At Week 12
  Percentage of participants achieving a histologic remission, defined as Geboes <2B at Week 12. Geboes is a grading system for histologic ulcerative colitis disease activity with scores ranging from 0 (no activity) to 5.4 (ulcer or granulation tissue).
Percentage of Participants with Histologic-Endoscopic Mucosal Improvement | At Week 12
  Percentage of participants achieving Geboes <= 3.1 and ES = 0 or 1 (normal appearance of mucosa or mild disease) at Week 12. Geboes is a grading system for histologic ulcerative colitis disease activity with scores ranging from 0 (no activity) to 5.4 (ulcer or granulation tissue).
Percentage of Participants with Histologic-Endoscopic Remission | At Week 12
  Percentage of participants achieving Geboes < 2 and ES = 0 or 1 (normal appearance of mucosa or mild disease) at Week 12. Geboes is a grading system for histologic ulcerative colitis disease activity with scores ranging from 0 (no activity) to 5.4 (ulcer or granulation tissue).
Percentage of Participants with Maintenance of Remission | Week 12 and Week 52
  Percentage of participants with clinical remission at both Week 12 and Week 52. Clinical remission is defined as mMS <= 2 with SFS = 0 or 1 (up to 1-2 stools more than normal), RBS = 0 (no blood seen) and ES = 0 or 1 (normal appearance of mucosa or mild disease). mMS is a composite score of ulcerative colitis disease activity, given by the sum of three subscores: SFS, RBS and ES. Each subscore is measured on a scale from 0 to 3, with higher values associated with greater severity.
Percentage of Participants with Corticosteroid-Free Remission | At Week 52
  Percentage of participants in clinical remission at Week 52 with no corticosteroid use at least 8 weeks prior to Week 52. Clinical remission is defined as mMS <= 2 with SFS = 0 or 1 (up to 1-2 stools more than normal), RBS = 0 (no blood seen) and ES = 0 or 1 (normal appearance of mucosa or mild disease). mMS is a composite score of ulcerative colitis disease activity, given by the sum of three subscores: SFS, RBS and ES. Each subscore is measured on a scale from 0 to 3, with higher values associated with greater severity.
Percentage of Participants with Endoscopic Improvement | At Week 52
  Percentage of participants achieving endoscopic subscore of 0 or 1 (normal appearance of mucosa or mild disease) at Week 52.
Percentage of Participants with Endoscopic Remission | At Week 52
  Percentage of participants achieving endoscopic subscore of 0 (normal appearance of mucosa) at Week 52.
Percentage of Participants with Histologic Improvement | At Week 52
  Percentage of participants achieving histologic improvement defined as Geboes <= 3.1 at Week 52.
Percentage of Participants with Histologic Remission | At Week 52
  Percentage of participants achieving histologic remission defined as Geboes <2B at Week 52.
Percentage of Participants with Histologic-Endoscopic Mucosal Improvement | At Week 52
  Percentage of participants achieving Geboes <= 3.1 and ES = 0 or 1 (normal appearance of mucosa or mild disease) at Week 52. Geboes is a grading system for histologic ulcerative colitis disease activity with scores ranging from 0 (no activity) to 5.4 (ulcer or granulation tissue).
Percentage of Participants with Histologic-Endoscopic Remission | At Week 52
  Percentage of participants achieving Geboes < 2 and ES = 0 or 1 (normal appearance of mucosa or mild disease) at Week 52. Geboes is a grading system for histologic ulcerative colitis disease activity with scores ranging from 0 (no activity) to 5.4 (ulcer or granulation tissue).
Percentage of Participants with Clinical remission: Among Biomarker-Defined Subgroups of Participants | At Week 12
  Percentage of participants achieving mMS <= 2 with SFS = 0 or 1 (up to 1-2 stools more than normal), RBS = 0 (no blood seen) and ES = 0 or 1 (normal appearance of mucosa or mild disease) at Week 12 in biomarker-defined subgroups. mMS is a composite score of ulcerative colitis disease activity, given by the sum of three subscores: SFS, RBS and ES. Each subscore is measured on a scale from 0 to 3, with higher values associated with greater severity.
Percentage of Participants with Clinical remission: Among Biomarker-Defined Subgroups of Participants | At Week 52
  Percentage of participants achieving mMS <= 2 with SFS = 0 or 1 (up to 1-2 stools more than normal), RBS = 0 (no blood seen) and ES = 0 or 1 (normal appearance of mucosa or mild disease) at Week 52 in biomarker-defined subgroups. mMS is a composite score of ulcerative colitis disease activity, given by the sum of three subscores: SFS, RBS and ES. Each subscore is measured on a scale from 0 to 3, with higher values associated with greater severity.
Percentage of Participants with Endoscopic Improvement: Among Biomarker-Defined Subgroups of Participants | At Week 12
  Percentage of participants achieving endoscopic subscore of 0 or 1 (normal appearance of mucosa or mild disease) at Week 12 in biomarker-defined subgroups.
Percentage of Participants with Endoscopic Improvement: Among Biomarker-Defined Subgroups of Participants | At Week 52
  Percentage of participants achieving endoscopic subscore of 0 or 1 (normal appearance of mucosa or mild disease) at Week 52 in biomarker-defined subgroups.
Change in Bowel Urgency | Baseline through Week 52
  Change in bowel urgency from baseline through Week 52. Bowel urgency is measured on a scale from 0 (None) to 4 (Severe).
Change in Abdominal Pain | Baseline through Week 52
  Change in abdominal pain from baseline through Week 52. Abdominal pain is measured on a scale from 0 (None) to 4 (Severe).
Change in Fatigue | Baseline to Week 12 and Week 52
  Change in fatigue as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) from baseline to Week 12 and Week 52. FACIT-Fatigue is a 13-item self-reported assessment of the level and impact of fatigue. The overall FACIT-Fatigue score ranges between 0 and 52, with higher scores associated with better quality of life concerns related to fatigue.
Change in Health-Related Quality of Life | Baseline to Week 12 and Week 52
  Change in Inflammatory Bowel Disease Questionnaire (IBDQ) score from baseline to Week 12 and Week 52. IBDQ is a 32-item self-reported assessment of health-related quality of life in participants with inflammatory bowel disease. The overall IBDQ score ranges from 32 to 224, with higher scores associated with better health-related quality of life.
Overall Change in UC Symptoms | Baseline to Week 2, Week 12, and Week 52
  Patient Global Impression of Change (PGIC) from baseline to Weeks 2, 12 and 52. PGIC measures overall change in ulcerative colitis symptoms from "Much better" to "Much worse".
Overall Severity in UC Symptoms | Baseline to Week 2, Week 12, and Week 52
  Patient Global Impression of Severity (PGIS) from baseline to Weeks 2, 12 and 52. PGIS measures severity of ulcerative colitis symptoms from "None" to "Very severe".
Incidence and Severity of Adverse Events (AEs) | Up to 70 Weeks after Baseline
  Incidence and severity of AEs, including serious AEs, AEs leading to treatment discontinuation and AEs of special interest.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (242):
- United States (90):
  - Digestive Health Specialists of the Southeast (Gastroenterology Associates of Dothan) - Dothan, Dothan, Alabama
  - Sun City Clinical Research, Glendale, Arizona
  - Arizona Digestive Health, P.C (ADH), Sun City, Arizona
  - University of Arizona-CATS Research Center, Tucson, Arizona
  - 310 Clinical Research, Inglewood, California
  - Om Research LLC, Lancaster, California
  - UCLA, Los Angeles, California
  - University of California Irvine, Orange, California
  - Stanford Medicine Outpatient Center, Redwood City, California
  - Acclaim Clinical Research, Inc., San Diego, California
  - Kaiser Permanente, San Francisco, California
  - UCSF/Medical Center at Mount Zion, San Francisco, California
  - Amicis Research Center, Santa Clarita, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Peak Gastroenterology Surgery Center, Lone Tree, Colorado
  - Access Research Institute, Brooksville, Florida
  - Gastro Florida, Clearwater, Florida
  - HealthMed Clinical Center Inc., Coral Gables, Florida
  - J&A Clinical Research, Doral, Florida
  - Clinical Research of Osceola, LLC, Kissimmee, Florida
  - Auzmer Research, Lakeland, Florida
  - Florida Research Institute - Lakewood, Lakewood Rch, Florida
  - Homestead Associates in Research, Inc., Miami, Florida
  - Allied Biomedical Research Institute, Inc, Miami, Florida
  - Miami Beach Clinical Research Center, Miami Beach, Florida
  - Eminat Research Group, Miramar, Florida
  - Orlando Regional Healthcare, Orlando, Florida
  - Nodal Medical Center, LLC, Tampa, Florida
  - Theia Clinical Research Centers, LLC, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Florida Medical Clinic, Zephyrhills, Florida
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Next Innovative Clinical Research, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Gastroenterology Health Partners, PLLC, New Albany, Indiana
  - Tri-State Gastroenterology Associates, Crestview Hills, Kentucky
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - Gastroenterology Health Partners, PLLC, Louisville, Kentucky
  - Louisiana Research Center - GastroIntestinal Associates, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Brigham & Womens Hosp, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, North Worcester, Massachusetts
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Allied Gastrointestinal Associates, PA, Flowood, Mississippi
  - Gastroenterology Associates and Endoscopy Center of North Mississippi, Oxford, Mississippi
  - BVL Clinical Research, Liberty, Missouri
  - Las Vegas Clinical Trials, LLC, North Las Vegas, Nevada
  - Intercity Gastroenterology, Fresh Meadows, New York
  - Northwell Health Physician Partners Gastroenterology at Great Neck, Great Neck, New York
  - Pioneer Clinical Research NY, New York, New York
  - New York-Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - Mainstreet - Richmond Hill Clinic, Richmond Hill, New York
  - Digestive Health Partners, PA, Asheville, North Carolina
  - Peters Medical Research (PMR), LLC, High Point, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Digestive Disease Consultants, Brunswick, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Gastroenterology Group, Columbus, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Gastro Intestinal Research Institute of Northern Ohio, Westlake, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - University Gastroenterology, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Gastro One, Cordova, Tennessee
  - Gastrointestinal Associates of Northeast Tennessee, Johnson City, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Texas Digestive Disease Consultants - Cedar Park, Cedar Park, Texas
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Proactive El Paso,LLC, El Paso, Texas
  - GI Alliance, Garland, Texas
  - Baylor College of Medicine., Houston, Texas
  - Integrity Advanced Therapeutics PLLC, Houston, Texas
  - TDDC dba GI Alliance Research, Mansfield, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - Digestive System Healthcare - Biopharma Informatic, LLC, Pasadena, Texas
  - Carta - Clinical Associates In Research Therapeutics Of America;LLC, San Antonio, Texas
  - Southern Star Research Institute, LLC., San Antonio, Texas
  - GI Alliance - Southlake, Southlake, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Tidewater Gastroenterology Pllc T/A Gastro. Assoc. of Tidewater, Chesapeake, Virginia
  - Gastroenterology Consultants and Endoscopy Center of Southwest Virginia, Roanoke, Virginia
  - The Vancouver Clinic, Vancouver, Washington
  - Marshall Health, Huntington, West Virginia
  - Univ of Wisconsin Hosp & Clin, Madison, Wisconsin
- Argentina (2):
  - CIPREC Centro de Investigacion y Prevencion Cardiovascular, Ciudad Autonoma Buenos Aires
  - Expertia S.A- Mautalen Salud e Investigación, Ciudad Autonoma Buenos Aires
- Australia (5):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Lyell McEwin Hospital, Adelaide, South Australia
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck
  - Barmherzige Brüder Wien, Vienna
  - Medizinische Universität Wien, Vienna
- Belgium (3):
  - AZ Maria Middelares, Ghent
  - CHC MontLégia, Liège
  - CHU de Liège (Sart Tilman), Liège
- Brazil (4):
  - Centro Digestivo de Curitiba, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre X, Porto Alegre, Rio Grande do Sul
  - CPQuali Pesquisa Clinica Ltda, São Paulo, São Paulo
  - BR Trials - Pesquisa Clínica, São Paulo, São Paulo
- MHAT St. Ivan Rilski, Gorna Oryahovitsa, Bulgaria
- South Edmonton Gastroenterology, Edmonton, Alberta, Canada
- Chile (3):
  - Hospital Guillermo Grant Benavente, Concepción
  - Clinica Universidad de Los Andes, Santiago
  - Medwal, Santiago
- China (23):
  - Peking University Third Hospital, Beijing
  - Binzhou Medical university hospital, Binzhou
  - the First Hospital of Jilin University, Changchun
  - Sichuan Provincial People's Hospital, Chengdu
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The sixth affiliated hospital of Sun Yat-Sen University, Guangzhou
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huizhou First Hospital, Huizhou
  - Jinhua municipal central hospital, Jinhua
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - Nanjing 1st Hospital, Nanjing
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Peking University Shenzhen Hospital, Shenzhen
  - Hebei Medical University - The Second Hospital, Shijiazhuang
  - Tianjin Medical University General Hospital, Tianjin
  - Wuhan Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Ren Min Hospital Affiliated Wu Han University, Wuhan
  - Wuxi People's Hospital, Wuxi
  - The Second Affiliated Hospital of Xi'an Jiao Tong University, Xi'an
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhuzhou Central Hospital, Zhuzhou
- Borzan Polyclinic, Osijek, Croatia
- Czechia (3):
  - SurGal Clinic s.r.o., Brno
  - Nemocnice Ceske Budejovice a.s., České Budějovice
  - Gastroenterologie s.r.o., Hradec Králové
- Herlev Hospital, Herlev, Denmark
- France (13):
  - CHU Amiens - Hopital Sud, Amiens
  - CHU Dijon Bourgogne Hôpital François Mitterand, Dijon
  - CH Dptal Les Oudairies, La Roche-sur-Yon
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - Hopital Nord, Marseille
  - Institut des MICI, Clinique Ambroise Paré, Neuilly-sur-Seine
  - CHU Nice - Hopital de l'Archet 2, Nice
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Robert Debre, Reims
  - CHU de Rennes - Hopital de Pontchaillo, Rennes
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - Hôpital de Rangueil, Toulouse
- Universitaetsklinikum Jena, Jena, Germany
- Hungary (6):
  - Clinexpert Kft., Budapest
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Clinexpert Gyongyos Kft, Gyöngyös
  - Clinfan Szolgaltato Kft., Szekszárd
  - Jávorszky Ödön Kórház, Vác
- India (3):
  - Surat Institute of Digestive Sciences Hospitals, Surat, Gujarat
  - Gujarat Gastro and Vascular Hospital, Surat, Gujarat
  - SR Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
- Shaare Zedek Medical Center, Jerusalem, Bayit Vegan, Israel
- Italy (5):
  - Ospedale Madonna delle Grazie, Matera, Basilicate
  - Universita'degli Studi di Napoli Federico II, Napoli, Campania
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Lombardy
  - ASST Rhodense - Ospedale di Rho, Rho, Lombardy
- Japan (19):
  - Tsujinaka Hospital Kashiwanoha, Chiba
  - Fukuoka University Hospital, Fukuoka
  - Hidaka Coloproctology Clinic, Fukuoka
  - Japanese Red Cross Takayama Hospital, Gifu
  - Aoyama Clinic;GI Endoscopy & IBD Center, Hyōgo
  - Kagawa Prefectural Central Hospital, Kagawa
  - Sameshima Hospital, Kagoshima
  - Gokeikai Ofuna Chuo Hospital, Kanagawa
  - Nagasaki University Hospital, Nagasaki
  - National Hospital Organization Osaka National Hospital, Osaka
  - Ishida Clinic of IBD and Gastroenterology, Ōita
  - Saga-ken Medical Centre Koseikan, Saga
  - Saga University Hospital, Saga
  - National Hospital Organization Shizuoka Medical Center, Shizuoka
  - Matsuda Hospital, Shizuoka
  - Kitasato University Kitasato Institute Hospital, Tokyo
  - JCHO Tokyo Yamate Medical Center, Tokyo
  - Tokai University Hachioji Hospital, Tokyo
  - Yokohama City University Medical Center, Yokohama
- Mexico (4):
  - Boca Clinical Trials Mexico S.C. (Guadalajara), Guadalajara, Jalisco
  - Accelerium S. de R.L. de C.V., Monterrey, Nuevo León
  - Hospital General de Mexico, Mexico, Tlaxcala
  - Medical Care & Research SA de CV, Mérida, Yucatán
- Poland (19):
  - SPZOZ w ??cznej, ??czna
  - Clinical Trials UMED Sp. z o. o., ?ód?
  - Centrum Medyczne "Medis", Bydgoszcz
  - Centrum Medyczne Lukamed Joanna Luka-Wendrowska, Chojnice
  - Endo-Med Sp. z o.o., Karczew
  - Allmedica Badania Kliniczne Sp z o.o. Sp K., Nowy Targ
  - Wojewodzki Specjalistyczny Szpital w Olsztynie, Olsztyn
  - NZOZ Eskulap Pabianice, Pabianice
  - Trialmed CRS, Piotrkow Trybunalski
  - SOLUMED Centrum Medyczne, Późna
  - Centrum Medyczne "MEDYK", Rzeszów
  - Kiepury Clinic, Sosnowiec
  - Gastromed Sp. z o.o., Toru?
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Vistamed & Vertigo Spó?Ka Z Ograniczon? Odpowiedzialno?Ci?, Wroc?aw
  - Penta Hospitals Polska, Wroc?aw
  - Melita Medical, Wroclaw
  - ETG Zamosc, Zamo??
- Portugal (6):
  - Hospital de Braga, Braga
  - Hospital da Luz Lisboa, Lisbon
  - Centro Hospitalar do Algarve - Hospital de Portimao, Portimão
  - Hospital de Sao Joao, Porto
  - Centro Hospitalar de Entre Douro e Vouga - H. São Sebastião, Santa Maria da Feira
  - Hospital Sao Teotonio, Viseu
- University of Puerto Rico - Medical Science Campus, San Juan, Puerto Rico
- Romania (2):
  - Colentina Clinical Hospital, Bucharest
  - Cantacuzino Clinical Hospital, Bucharest
- Serbia (6):
  - University Hospital Center Dr Dragisa Misovic - Dedinje, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - University Hospital Medical Center Bezanijska Kosa, Belgrade
  - University Hospital Medical Center Zvezdara, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Vojvodina, Novi Sad
- Slovakia (2):
  - Cliniq s.r.o., Bratislava
  - Endomed, s.r.o., Košice
- Spain (2):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Taiwan (3):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua, Changhua County
  - National Taiwan University Hospital, Taipei, Zhongzheng District
  - E-Da Hospital, Kaohsiung City
- Thailand (6):
  - Division of Gastroenterology, Depart of Medicine, Fac of Med., Chulalongkorn University, Bangkok
  - Division of Gastroenterology, Depart of Internal Med, Siriraj H, Mahidol Uni, Bangkok
  - Liver Research Unit, Srinagarind Hospital, Khon Kaen
  - Thammasat University Hospital, Pathum Thani
  - Division of Gastroenterology, Depart of Medicine, Fac. of Med, Songklanagarind University, Songkhla
  - Surin hospital, Surin
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge
  - Royal Liverpool University Hospital, Liverpool
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing